CLINICAL TRIAL: NCT05688007
Title: The Association Between Parathyroid Hormone and Preterm Labor
Status: Completed | Type: Observational
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Rania Hassan Mostafa, Principal Investigator, Ain Shams Maternity Hospital
Other Study IDs: MS 168/2021
Record Dates: First submitted 2023-01-09; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Preterm Labor; Parathyroid Diseases
Keywords: parathyroid hormone; calcium, magnesium, phosphorus, albumin
MeSH Terms: conditions — Obstetric Labor, Premature; Parathyroid Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: pregnant women with established preterm labor - gestational age: (28-36 weeks), having: Regular uterine contractions are at least 3 in 10 min each lasting 40 seconds. Progressive cervical dilatation (at least 4 cm).
  Interventions: Diagnostic Test: parathyroid hormone level; Diagnostic Test: serum electrolytes
- Controls: pregnant women not in labor - gestational age: (28- 36 weeks)
  Interventions: Diagnostic Test: parathyroid hormone level; Diagnostic Test: serum electrolytes

INTERVENTIONS:
Diagnostic Test: parathyroid hormone level — Serum level of parathyroid hormone
Diagnostic Test: serum electrolytes — Serum levels of: magnesium, phosphorus, calcium, and albumin

SUMMARY:
This observational study aims to test the level of parathyroid hormone in pregnant women. The main question it aims to answer is:

n Pregnant women, are the levels of serum PTH, calcium, magnesium, phosphorus & albumin similar in both preterm and term births?

DETAILED DESCRIPTION:
* Approval from ethical committee will be sought.
* Patients will be enrolled from Ain Shams University Maternity Hospital labor ward and antenatal outpatient clinic.
* History, examination and fetal ultrasound will be done to identify eligible patients.

History: a full detailed history including personal, menstrual, obstetric, present, past history and family history will be obtained.

Accurate last menstrual period date will be obtained, and gestational age will be calculated using Naegele's rule or first trimester ultrasound to identify preterm patients with gestational age (28-36 weeks).

Examination: general, abdominal and vaginal examination to identify patients in established labor with Regular uterine contractions are at least 3 in 10 min each lasting 40 seconds. Progressive cervical dilatation (at least 4 cm). Ultrasound: for (viability of fetus, fetal biometry and estimated fetal weight, amniotic fluid, placental localization).

Thus, two groups of patients will be identified:

1. Cases: established preterm labor - gestational age: (28-36 weeks)
2. Controls: pregnant women not in labor - gestational age: (28- 36 weeks)

   * Venous blood samples will be withdrawn about (3ml) once from every patient within one hour from inclusion into the study to measure serum parathyroid hormone, calcium, magnesium, phosphorus and albumin levels.
   * Samples will not be collected from an arm with an intravenous catheter if alternate sites are available.
   * Patient collection site will be appropriately disinfected prior to sample collection.
   * After collection, samples will be put in a red or yellow tube (serum separating tube) with a serum gel separator.
   * Samples will be gently mixed immediately following collection into tube to ensure proper preservation of the analytes. 180° tube inversion, allowing bubble to travel the length of the tube, followed by return to upright position is one mix.
   * Samples will be delivered to laboratory within 30 to 60 minutes.
   * Data will be collected and recorded in a case report form (Age, parity, previous preterm births/ miscarriage, gestational age, measured levels of serum PTH, calcium, magnesium, phosphorus & albumin , mode of delivery, birth weight).
   * Statistical analysis will be done to get results.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged (18-40).
* Gestational age (28-36 weeks).

Exclusion Criteria:

* Known maternal disease as diabetes, hypertension, renal disease, cardiac disease and liver disease.
* Known hypo or hyperparathyroidism
* Multiple pregnancy
* Polyhydramnios
* Premature rupture of membrane
* Antepartum Hemorrhage
* Uterine malformations e.g. bicornuate uterus
* Smoking

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women attending Ain Shams University Maternity Hospital (labor ward and antenatal outpatient clinic)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-10-16 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
parathyroid hormone | 1 day
  serum level of parathyroid hormone (ng/L)

SECONDARY OUTCOMES:
Calcium | 1 day
  serum calcium level (mg/dl)
Magnesium | 1 day
  serum magnesium level (meq/L)
Phosphorus | 1 day
  serum phosphorus level (mg/dl)
Albumin | 1 day
  serum albumin level (g/dl)

CONTACTS AND LOCATIONS:
Overall Officials: Sherif A Ashoush, MD, Study Director — Faculty of Medicine Ain Shams University
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
protocol and dataset (analytic code) can be sent via email upon reasonable requests
Supporting Information: Study Protocol, Analytic Code
Time Frame: after publication of the manuscript, and for one year after.
Access Criteria: via email (raneyah@gmail.com)